CLINICAL TRIAL: NCT05257512
Title: A Phase I/II, Open-label, Multicenter Study of the Safety, Pharmacokinetics, and Antitumor Activity of SY-3505 Capsule in Patients With ALK-positive Advanced Non-small Cell Lung Cancer
Brief Title: Phase I/II Study of SY-3505 in Patients With ALK-positive Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-3505-I
Record Dates: First submitted 2022-02-09; First posted 2022-02-25 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: SY-3505; ALK; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I/II Study of SY-3505 (Experimental): SY-3505 will be given orally in ascending doses (escalation cohort), until the DLT or RP2D is reached. Up to 6 patients will then be enrolled in the expansion cohort at the recommended dose. In phase II, SY-3505 will be given at RP2D in advanced ALK-positive NSCLC patients.
  Interventions: Drug: SY-3505

INTERVENTIONS:
Drug: SY-3505 — The third-generation ALK TKI
  Other Names: CT-3505

SUMMARY:
This is a phase I/II, open-label and multi-center study of SY-3505, a third-generation ALK TKI, in patients with advanced ALK-positive non-small cell lung cancer (ALK-positive NSCLC).

DETAILED DESCRIPTION:
The study consists of two parts:

Part 1: Dose-escalation and dose-expansion in patients with advanced ALK-positive NSCLC, including 9 SY-3505 dose levels.

Dose-escalation study phase is designed to determine the dose-limiting toxicity (DLT) according to a 3+3 design and recommended phase II dose (RP2D) and to characterize the safety, tolerability, and pharmacokinetics (PK) profile of SY-3505. Other dose regimens may be explored based on the analysis of emerging PK and safety data. At this study phase, SY-3505 administered orally once daily (QD) in 28-day treatment cycles to adult patients with ALK-positive NSCLC. Dose-expansion study is designed to evaluate the antitumor activity (ORR, DCR and DoR) of SY-3505 at selected doses in ALK-positive NSCLC patients who have received at least 1 prior ALK TKI therapy.

Part 2: Phase 2 study to evaluate the efficacy of SY-3505.

This phase is designed to determine the antitumor activity (ORR, DCR, DoR, PFS and OS), safety, and PK of SY-3505 at RP2D in ALK-positive NSCLC patients who have received alectinib only or ≥2 prior ALK TKIs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years at the time of screening.
2. Must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
3. Estimated Life expectancy ≥ 12 weeks.
4. Must have either at least one measurable lesion with no prior local treatment or measurable lesions with definite progression (Bone metastases alone were not accepted) after local treatment per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Dose-escalation phase: patients must have histological or cytological confirmed ALK-positive advanced NSCLC. Dose-expansion phase: patients must have histological or cytological confirmed ALK-positive advanced NSCLC and progressed after at least one prior line of ALK TKI therapy. Phase II: patients must have histological or cytological confirmed ALK-positive advanced NSCLC and progressed after only alectinib or ≥2 prior ALK TKIs treatment. The pathological report requires either positivity for ALK gene expression determined by fluorescence in-situ hybridization (FISH) assay, immunohistochemistry (IHC), reverse transcription-polymerase chain reaction (RT-PCR), next-generation sequencing (NGS) or other identified methods from previous reports and provide tissue for ALK retest if possible or providing tissue for ALK test if no previous report is available.
6. Patients without brain metastasis or with asymptomatic brain metastases (no need for intervention or stable more than 4 weeks after treated).
7. Adequate organ function within 10 days prior to the study of treatment as defined in the below:

   Hepatic function

   Total serum bilirubin (TBIL) ≤ 1.5 times upper limit of normal (ULN); Aspartate transaminase (AST), alanine transaminase (ALT) and γ- glutamyltransferase (GGT) ≤ 2.5 times ULN if no demonstrable liver metastases, or otherwise ≤ 5 times ULN.

   Bone marrow function

   Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L; Platelets (PLT) count ≥ 100 x 10⁹/L; Hemoglobin (Hb) ≥ 90 g/L.

   Renal function

   Creatinine clearance ≥ 60 mL/min.

   Pancreatic function

   Serum total amylase ≤1.5 times ULN; Serum lipase ≤ 1.5 times ULN.

   Blood glucose

   Fasting Blood Glucose (FBG) ≤ 200 mg/dL (11.1 mmol/L).

   Serum lipid

   Serum cholesterol ≤ 500 mg/dL (12.92 mmol/L).

   Cardiac function

   Left ventricular ejection fraction (LVEF) ≥ 50%.
8. Any toxicity of previous antineoplastic treatments was restored to ≤ 1 (except hair loss).
9. Female patients with reproductive potential must have a negative serum pregnancy test, male and female patients of childbearing potential must be willing to completely abstain or agree to use an appropriate method of contraception during the entire study duration and for at least 3 months after the last dose of study medication.
10. Willingness and ability to give informed consent and follow protocol procedures, and comply with follow-up visit requirements.

Exclusion Criteria:

1. Any of the following within 6 months prior to starting trial treatment: Cerebrovascular accident/ stroke, myocardial infarction, severe/ unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), second- or third- degree atrioventricular (AV) block (unless paced) or any AV block with PR interval >220 msec, or any grade of uncontrolled atrial fibrillation.
2. ECG evaluated QT interval corrected (Fridericia) (QTcF) of > 450 msec in males or > 470 msec in females or congenital long QT syndrome.
3. Grade ≥ 3 peripheral neuropathy (CTCAE version 5.0).
4. Any active autoimmune diseases or history of autoimmune diseases that require long-term steroid or other immunosuppressants treatment.
5. Previous medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
6. Patients being treated with any anticoagulants, prone to bleeding, or have a coagulation disorder.
7. Active hepatitis (Hepatitis B: HBsAg-positive and HBV-DNA ≥ 2000 IU/ mL; Hepatitis B: HCV antibody-positive and HCV-RNA ≥ 1000 IU/ml), HIV antibody-positive; Active syphilis.
8. Patient underwent major surgery within 4 weeks prior to starting trial treatment.
9. Patients received radical radiotherapy within 4 weeks, palliative radiotherapy within 2 weeks, or radioactive agents (strontium, samarium, etc.) within 8 weeks prior to starting trial treatment.
10. Patients received systemic antitumor therapy, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokine or cancer growth control factor), or clearly indicated antitumor traditional Chinese medicine within 4 weeks (targeted therapy within 2 weeks) prior to starting trial treatment.
11. Patients treated with the following drugs and could not be discontinued at least 7 days prior to starting trial treatment and during the entire study duration: drugs known to be strong inducers or suppressors of CYP3A (for details, see prohibited combination drugs in this trial).
12. Patients with any active infection requiring systemic therapy within 4 weeks prior to starting trial treatment.
13. Comorbidities that may seriously endanger the patient's safety or affect the completion of the trial, such as severe diabetes, according to the judgment of investigator.
14. A clear previous history of neurological or psychiatric disorders, including dementia or diagnosed epilepsy for any reason.
15. With a history (within 5 years) or presence of other malignancies, excluding cured skin basal cell carcinoma and carcinoma in situ of the cervix.
16. Other situations that may increase the risks related to the study medication, interfere with the interpretation of the study results, affect compliance of the trial, etc. are determined by the investigator to be not suitable for the trial.
17. In phase II: previously received third-generation ALK TKIs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-04-26 (Actual); Primary Completion 2024-04-26 (Estimated); Study Completion 2024-08-26 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence rate of dose limiting toxicities (DLTs) during the first cycle of treatment | Dose-escalation Cycle 1 (each cycle is 28 days)
  Maximum Tolerated Dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) in Cycle 1.
Phase I: Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
  Characterization of the safety and tolerability
Phase II: Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Anti-tumor activity of SY-3505

SECONDARY OUTCOMES:
Phase I: Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary anti-tumor activity of SY-3505
Phase I & II: Disease control rate (DCR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary anti-tumor activity of SY-3505
Phase I & II: Duration of response (DOR) | Up to 24 months
  Anti-tumor activity of SY-3505
Phase I & II: Progression-free survival (PFS) | Up to 24 months
  Anti-tumor activity of SY-3505
Phase I & II: Overall survival (OS) | Up to 24 months
  Anti-tumor activity of SY-3505
Phase I & II: Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
  Characterization of the safety and tolerability
Phase I & II: Pharmacokinetics (Cmax) for SY-3505 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as maximum observed plasma concentration
Phase I & II: Pharmacokinetics (Tmax) for SY-3505 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as time to maximum plasma concentration
Phase I & II: Pharmacokinetics (AUC0-t) for SY-3505 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Phase I & II: Pharmacokinetics (t½) for SY-3505 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as the apparent plasma terminal phase disposition half-life
Phase I & II: Pharmacokinetics (Cl/F) for SY-3505 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as oral dose clearance

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Hu X, Li X, Gong C, Wang K, Li Y, Zhang S, Luo Y, Wang P, Jiang L, Meng X, Dong X, Wang H, Yang R, Mei Q, Liu B, Yang L, Sun Y. Ficonalkib (SY-3505) in Advanced ALK-Positive NSCLC: A Multicenter, Open-Label, Single-Arm, Phase 1/2 Study. J Thorac Oncol. 2024 Jun;19(6):898-911. doi: 10.1016/j.jtho.2024.01.015. Epub 2024 Jan 29. PMID 38295954